CLINICAL TRIAL: NCT03966625
Title: Serological Identification of Celiac Disease in Kids (Swedish: Screening för Celiaki på Barnmottagning)
Brief Title: Serological Identification of Celiac Disease in Kids
Acronym: SICK
Status: Completed | Type: Observational
Sponsor: Sahlgrenska University Hospital (Other)
Collaborators: Vastra Gotaland Region (Other Government)
Responsible Party: Principal Investigator, Karl Mårild, Pediatrican, associate professor, Sahlgrenska University Hospital
Other Study IDs: DSBUS
Record Dates: First submitted 2019-05-25; First posted 2019-05-29 (Actual); Last update posted 2021-12-09 (Actual); Status verified 2021-12

CONDITIONS: Celiac Disease in Children; Pediatric Disorder; Health, Subjective; Growth Delay
Keywords: screening

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: tissue transglutaminase autoantibodies — celiac disease-specific autoantibodies

SUMMARY:
The investigators aim to examine the feasibility of incorporating serological celiac disease (CD) screening into general pediatric outpatient clinics in Sweden and through structured monitoring examine the effects of diagnosing and treating screening-detected CD.

Screening will be tailored to general pediatric outpatient clinics in the Gothenburg metropolitan area with the goal to screen 1000 children over four months. Screening for CD will be carried out by measuring tissue transglutaminase autoantibodies (TGA) in blood. Children who are persistently TGA positive will be enrolled into a 6-12-month follow-up protocol responsible for diagnosing CD, installation of gluten-free diet and to assess their short-term impact upon the child's wellbeing. Other components to assess include (I) the feasibility to incorporate CD screening into busy pediatric practices; (II) parental/child interest in, and satisfaction with, participating in a CD screening program and (III) identifying key considerations for a possible scaled-up, broad-based, CD screening.

ELIGIBILITY:
Inclusion Criteria:

* Aged 2-17 years old
* Patient at pediatric outpatient clinics in Gothenburg metro area
* Parental and adolescent consent to screening

Exclusion Criteria for serological screening:

* Established celiac disease diagnosis
* Type 1 diabetes

Ages: 2 Years to 17 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: Patients at pediatric outpatient clinics in Gothenburg metro area
Sampling Method: Non-Probability Sample
Enrollment: 496 (Actual)
Dates: Start 2019-11-04 (Actual); Primary Completion 2021-07-01 (Actual); Study Completion 2021-07-01 (Actual)

PRIMARY OUTCOMES:
Number of participants diagnosed with celiac disease | Assessed after 6-12 months of follow-up
  Celiac disease diagnosed according to European pediatric (ESPGHAN) guidelines

SECONDARY OUTCOMES:
Number of participants identified with celiac disease autoimmunity | Assessed after performed two tests of TTG (apprx. 1-2 months after enrollment)
  Celiac disease autoimmunity defined by having two consecutive positive tests for tissue transglutaminase (TTG) autoantibodies

CONTACTS AND LOCATIONS:
Locations (2):
- Sweden (2):
  - Queen Slivia Children's Hosptial, Gothenburg
  - BUMM Hisingen, Gothenburg

IPD SHARING:
Plan to Share IPD: No
Individual participant data will not be shared in accordance with the ethical approval of this study